CLINICAL TRIAL: NCT02078050
Title: Volontary Inspiratory Muscles Measures Compared With Phrenic Nerves Magnetic Stimulations Measures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2013-A00638-37
Record Dates: First submitted 2013-12-20; First posted 2014-03-05 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-02

CONDITIONS: Neuromuscular Diseases; Respiratory Failure
MeSH Terms: conditions — Neuromuscular Diseases; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phrenic nerves magnetic stimulations (Other)
  Interventions: Other: Phrenic nerves magnetic stimulations

INTERVENTIONS:
Other: Phrenic nerves magnetic stimulations

SUMMARY:
Respiratory failure is the main death cause in neuromuscular diseases. Non-invasive and volitional measures of inspiratory muscles strength include the nasal pressure with an occluded nostril (Psnip) and the maximal inspiratory pressure (PImax). Unfortunately, volitional maneuvers depend of patient effort. The aim of this research is to validate a non-invasive and non-volitional technique to evaluate diaphragm strength at neuromuscular diseases patients. The methodology consists to add to PImax and Psnip measures 5 phrenic nerves magnetical stimulation maneuvers (Pstim).Stimulations will be realize at 3 inspiratory pression levels (0, -1 cm H2O and -5 cm H2O).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and more men or women
* neuromuscular diseases
* Pimax and Snip evaluation Indication

Exclusion Criteria:

* pregnant women
* Usual contre-indications for nuclear magnetic resonance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Magnetic stimulation pressure measure (Pstim), according to 3 conditions : Pstime, Pstim-5 and Pstim-1 (measured in cmH20). The condition which is most correlated with maximal inspiratory pressure (Pimax or Psnip) is selected. | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital R. Poincaré, Garches, France